CLINICAL TRIAL: NCT01030796
Title: Quitting Caffeine for Better Glucose Metabolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: James D. Lane, Ph.D., Professor, Duke University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011009 (completed); R01DK067486 (NIH)
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Caffeine abstinence — Brief instruction on beginning and maintaining caffeine abstinence.

SUMMARY:
This project is a pilot study of caffeine abstinence in coffee-drinkers who have type 2 diabetes. Evidence suggests that caffeine may impair the control of glucose levels, especially in those people who have type 2 diabetes. Eliminating caffeinated beverages from the diet might improve glucose control, but the difficulty of quitting is unknown. This pilot study will follow a small number of type 2 diabetic patients for three months after a brief intervention designed to help people quit caffeine. Data on success with maintaining abstinence and on changes in glucose control will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 6-month history of type 2 diabetes
* impaired chronic glucose control (HbA1c >= 7%)
* daily consumption of 250 mg caffeine or more in coffee, tea, and other caffeinated beverages

Exclusion Criteria:

* use of exogenous insulin
* use of non-diabetes medications that impact glucose metabolism
* medical of psychiatric history that prevents participation or increases risk
* current pregnancy
* current participation in other clinical trials
* deemed unable to comply with the study protocol for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Caffeine abstinence | baseline, 2 weeks, 1, 2, and 3 months

SECONDARY OUTCOMES:
HbA1c | Baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James D Lane, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States